CLINICAL TRIAL: NCT03303066
Title: A Phase 2/3 Trial of FG-4592 for Treatment of Anemia in Subjects With Lower Risk Myelodysplastic Syndrome
Brief Title: Efficacy and Safety of FG-4592 for Treatment of Anemia in Participants With Lower Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FGCL-4592-813
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Anemia; Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndromes; Anemia; Hemoglobin (Hb); Low Risk Myelodysplastic Syndrome
MeSH Terms: conditions — Anemia; Myelodysplastic Syndromes | interventions — roxadustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Phase 2 part is an open label, single arm, dose-escalation study. Phase 3 component is a randomized, double blind, placebo-controlled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 2 Part: FG-4592 (Experimental): Fixed starting doses (different doses for lower body weight & higher body weight) of FG-4592 administered orally 3 times a week (TIW) for up to 26 weeks; dose adjustments to Hb levels are allowed during the study.
  Interventions: Drug: FG-4592
- Phase 3 Part: FG-4592 (Experimental): Fixed starting doses (different doses for lower body weight & higher body weight) of FG-4592 administered orally TIW for up to 26 weeks; dose adjustments to Hb levels are allowed during the study.
  Interventions: Drug: FG-4592
- Phase 3 Part: Placebo (Placebo Comparator): Placebo (matching to FG-4592) administered orally TIW for up to 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FG-4592 — Oral
  Other Names: Roxadustat; AZD9941
  Arms: Phase 2 Part: FG-4592; Phase 3 Part: FG-4592
Drug: Placebo — Oral
  Arms: Phase 3 Part: Placebo

SUMMARY:
The objective of this study to evaluate the efficacy FG-4592 for the treatment of anemia in Chinese participants with lower risk MDS.

DETAILED DESCRIPTION:
This is a Phase 2/3 trial with sequential Phase 2 and Phase 3 components. In each part, there is an up to 4 weeks screening period followed by a treatment period of 26 weeks and a 4 week follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of primary MDS classified as very low, low or intermediate risk with <5% blasts (documented within 12 weeks prior to Day 1)
* Screening Hb <10 g/dL and ≥6g/dL
* Transfusion independent defined as no red blood cell transfusions within 12 weeks of Day 1
* Erythropoiesis-stimulating agent (ESA)-naïve (not within 30 days of Day 1)
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2

Key Exclusion Criteria:

* Diagnosis of secondary MDS
* Significant myelofibrosis (>2+fibrosis)
* Prior therapy with azacitidine, decitabine, antithymocyte globulin, cyclosporine, thalidomide, or lenalidomide within 12 weeks prior to Day 1
* Baseline erythropoietin level of >400 units (U)/liter (L)
* Clinically significant anemia due to non-MDS etiologies

Note: Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With a Hemoglobin (Hb) Response to FG-4592 Without Transfusion | 26 weeks
  Hemoglobin response to FG-4592 is defined as an increase in mean Hb of ≥1.0 grams (g)/deciliter (dL) from baseline within any 8-week period during the study without transfusion.

SECONDARY OUTCOMES:
Number of Participants With Hb Increase ≥1.0 g/dL From Baseline | 26 weeks
  Hb response to FG-4592 is defined as an increase in mean Hb of ≥1.0 g/dL from baseline within any 8-week period during the study without transfusion.
Time to First Hb Response | 26 weeks
  Hb response to FG-4592 is defined as an increase in mean Hb of ≥1.0 g/dL from baseline within any 8-week period during the study without transfusion.
Change From Baseline in Mean Hb in Weeks 25 to 27 | Baseline, Weeks 25 to 27
Percentage of Participants With Mean Hb ≥10.0 g/dL Within Any 8-week Period During the Study Without Transfusion | 26 weeks
Number of Participants that Require Transfusions or Hb <6 g/dL up to Week 27 | Up to Week 27
Mean Change From Baseline in Functional Assessment of Cancer Therapy - Anemia (FACT-An) and Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Scores at Week 27 | 30 weeks
  Frame: Baseline, Week 27

CONTACTS AND LOCATIONS:
Locations (38):
- China (38):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Xiyuan Hospital, CACMS, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Nan Fang Hospital, Guangzhou, Guangdong
  - Zhuzhou Central Hospital, Zhuzhou, Guangdong
  - Hainan Central Hospital, Haikou, Hainan
  - Second hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tumor Hospital of Henan province, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Union Hospital Affiliated Tongji Medical College Huazhong University of Science and Technolog, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital Of Soochow University, Suzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Xuzhou Medical University, Jinan, Shandong
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tongji Hospital, Shanghai, Shanghai Municipality
  - Shaanxi Provincial People's Hospital, Xian, Shanxi
  - The First Affiliated Hospital of Xi'an Jiao Tong University Medical College, Xian, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Blood disease hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University Medical College, Hangzhou, Zhejiang